CLINICAL TRIAL: NCT05328336
Title: A Single-arm, Multicenter, Open Clinical Trial of the Efficacy and Safety of Tislelizumab in Combination With Nab-Paclitaxel for the Perioperative Treatment of Muscle-invasive Bladder Cancer
Brief Title: Perioperative Tislelizumab Combined With Nab-Paclitaxel for Muscle-invasive Urothelial Bladder Cancer: A Multicenter Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRUCE-11
Record Dates: First submitted 2022-04-06; First posted 2022-04-14 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-04

CONDITIONS: Muscle Invasive Bladder Cancer Urothelial Carcinoma
Keywords: neoadjuvant treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Tislelizumab and Nab Paclitaxel (Experimental): Experimental: Tislelizumab and Nab Paclitaxel Tislelizumab 200mg IV on day 1 in combination with nab paclitaxel 200mg IV on day 2 every 3 weeks for 3 cycles followed by surgery.
  Interventions: Drug: Tislelizumab Nab paclitaxel

INTERVENTIONS:
Drug: Tislelizumab Nab paclitaxel — Drug: Tislelizumab Tislelizumab 200mg will be administered on Day 1 every 3 weeks for 3 cycles
  Other Names:
  • BGB-A317 Drug: Nab paclitaxel Nab paclitaxel 200mg will

SUMMARY:
This is a single-arm, open-label, multicenter clinical trial to investigate the safety and efficacy of tislelizumab when given in combination with nab-paclitaxel as perioperative treatment in patients with muscle-invasive bladder cancer (MIBC) prior to cystectomy or complete TURBT. Patients will receive perioperative treatment with tislelizumab in combination with nab-paclitaxel every 3 weeks for 3 treatment cycles over 9 weeks followed by radical cystectomy or complete TURBT.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Ability to comply with the protocol.
3. Age ≥ 18 years.
4. Suitable and planned for complete transurethral resection of bladder tumor or radical cystectomy
5. At least one measurable lesion meeting RECISTv1.1 criteria prior to transurethral bladder tumor electrosurgery (MR/CT long diameter of ≥10 mm or short diameter of ≥15 mm of enlarged lymph node required for this measurable lesion according to RECISTv1.1)
6. Histopathologically confirmed urothelial carcinoma. Patients with mixed histologies are required to have a dominant (i.e. 50% at least) urothelial cell pattern.
7. Clinical stage T2-T4a NxM0 disease by CT (or MRI).
8. Expected survival time is greater than 12 weeks.
9. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 1 or 2.
10. Agree to provide tissue examination specimens (used to detect PD-L1 expression, tumor mutation burden, etc.)
11. The organ function level must meet the following requirements:

    * Hematological indicators: absolute neutrophil count ≥1.5×10^9/ L, platelet count ≥80×10^9/L, hemoglobin ≥6.0 g/dL (can be maintained by symptomatic treatment);
    * Liver function: total bilirubin ≤ 1.5 times the upper limit of normal value, alanine aminotransferase and aspartate aminotransferase

      ≤ 2.5 times the upper limit of normal value, if there is intrahepatic transaminase ≤ 5 times the upper limit of normal value;
    * Renal function: creatinine ≤ 2 times the upper limit of normal, and creatinine clearance ≥ 30 ml/min;

Exclusion Criteria:

1. Receive live attenuated vaccines within 4 weeks before treatment or plan to receive live attenuated vaccines during the study period.
2. Active, known or suspected autoimmune diseases.
3. Known history of primary immunodeficiency.
4. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
5. Female patients who are pregnant or breastfeeding.
6. Untreated acute or chronic active hepatitis B or C infection. In the case of patients receiving antiviral therapy, the doctor will judge whether they are eligible for enrollment according to the individual conditions of the patient while monitoring the virus copy number.
7. Have used immunosuppressive drugs in the past 4 weeks before starting treatment, excluding nasal spray and inhaled corticosteroids or physiological doses of systemic steroids (that is, prednisolone or equivalent physiological doses of no more than 10 mg/day) Other corticosteroids).
8. Those who are known or suspected to be allergic to tislelizumab and nab paclitaxel.
9. Have a clear history of active tuberculosis.
10. Have received PD-1/PD-L1/CTLA-4 antibody or other immunotherapy in the past.
11. Those who are participating in other clinical research.
12. Reproductive men or women who are likely to become pregnant have not taken reliable contraceptive measures.
13. Uncontrolled concurrent diseases include but are not limited to:

    * HIV-infected persons (HIV antibody positive).
    * Serious infections that are active or poorly clinically controlled.
    * There are serious or uncontrollable systemic diseases (such as severe mental, neurological, epilepsy or dementia, unstable or uncompensated respiratory, cardiovascular, liver or kidney diseases, uncontrolled hypertension [ie refers to After drug treatment, it is still greater than or equal to CTCAE Grade 2 hypertension]) evidence.
    * Active bleeding or new thrombotic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
complete response (CR) rate | At the time of complete transurethral resection of bladder tumor or radical cystectomy (within 12 weeks of the first dose of tislelizumab)
  defined as the percentage of participants having CR. CR is defined as absence of viable tumor in examined tissue

SECONDARY OUTCOMES:
Number of subjects that reach pathological downstaging to <pT2 | At the time of complete transurethral resection of bladder tumor or radical cystectomy (within 12 weeks of the first dose of tislelizumab)
  defined as pT0-T1N0M0 at the time of cystectomy or cTURBT
Objective response rate (ORR) | At the time of complete transurethral resection of bladder tumor or radical cystectomy (within 12 weeks of the first dose of tislelizumab)
  defined as the proportion of patients who have a partial or complete response to therapy
Event-free survival (EFS) | up to 3 years
  defined from D1 of neoadjuvant treatment until progression (in those who progress prior to surgery) or until recurrence (post-surgery) or until death as a result of any cause.
Overall Survival (OS) | up to 3 years
  defined as the number of days from study entry to death. Individuals who are alive at last contact will be censored on the date of last contact.
Number of adverse events and severity by grade (CTCAE) | up to 1 years
  Safety and toxicity will be characterized according to the reported adverse event (AE) profile using NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0, as well as a patient questionnaire derived from the Patient Reported Outcomes (PRO)-CTCAE and Patient Reported Outcomes Measurement Information System (PROMIS).

CONTACTS AND LOCATIONS:
Locations (1):
- ianjin Medical University Second Hospital, Tianjin, Tianjin Municipality, China